CLINICAL TRIAL: NCT02455531
Title: Long-term Outcomes of Children With HLHS (Hypoplastic Left Heart Syndrome) and the Impact of Norwood Shunt Type (A Study Conducted by the Pediatric Heart Network)
Brief Title: Long-term Outcomes of Children With Hypoplastic Left Heart Syndrome and the Impact of Norwood Shunt Type
Acronym: SVRIII
Status: Active, not recruiting | Type: Observational
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: U10HL068270-4b; U10HL068270 (NIH)
Record Dates: First submitted 2015-05-22; First posted 2015-05-28 (Estimated); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-03

CONDITIONS: Heart Defects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants and their parents who have not yet contributed to the SVR Extension biorepository will be offered the opportunity to provide saliva for extraction and storage of DNA. If study participants have consented to participate in the biorepository through the SVR Extension study but not yet contributed a sample, they will be asked to contribute at the time of the SVR III participation. Families who were not previously approached, or who declined participation in the biorepository earlier, may be offered the opportunity to participate at the time of the SVR III participation.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Transplant-free survivors: Transplant-free survivors of the SVR cohort (All SVR survivors are eligible to be followed for vital status.)

SUMMARY:
The purpose of this study is to compare direct and indirect measures of right ventricular (RV) systolic and diastolic function between 11 year old subjects who had been randomly assigned to receive a right ventricle to pulmonary artery shunt (RVPAS) vs. a modified Blalock-Taussig shunt (MBTS) at the time of the Norwood operation.

DETAILED DESCRIPTION:
The Single Ventricle Reconstruction (SVR) trial was the first multicenter, randomized clinical trial to compare two operations in the field of congenital heart disease.8,11 Children with HLHS and other related single RV lesions were enrolled and randomized to receive either a MBTS or a RVPAS at the time of the initial Norwood procedure. This landmark study provided extraordinary insight not only into the consequences of both shunt types, but also into the course, treatment responses and short- and mid-term outcomes for these medically complex patients. Through the SVR Trial and SVR Extension Study (SVR II), outcomes, including but not limited to the primary outcome of transplant-free survival, have now been evaluated in this patient cohort when the last enrolled patient reached 12 months and again at 3 years of age. While early post-operative transplant-free survival during the interstage period7 and at one year8 was better for those children randomized to a RVPAS, survival by the 3-year evaluation appeared equivalent between the two shunt types. Moreover, RVEF was somewhat diminished and the number of interventions was higher in the RVPAS group.12 These findings raised concern that the RV dysfunction in the RVPAS group may be progressive, leading to significantly worse long-term outcomes; if so, the benefits of the RVPAS for short-term survival may be outweighed by longer-term morbidity and mortality. Thus, the optimal surgical approach for newborns with HLHS and related single RV lesions remains unclear.

The Pediatric Heart Network (PHN) Investigators have a unique opportunity and responsibility to analyze the effect of the type of systemic-to-pulmonary artery shunt placed during the Norwood procedure on longer-term survival, as well as to define its effect on other long-term outcomes in this multi-institutional cohort of exquisitely characterized subjects with single RV lesions. As subjects enrolled in the SVR cohort approach a decade of age, the investigators aim: 1) to determine if shunt type at the time of Norwood operation is associated with any long-term differences in cardiac function, survival, or contributors to quality of life; and 2) to characterize long-term outcomes and determine risk factors other than shunt type for adverse long-term outcomes in children with HLHS and other related single ventricle anomalies.

ELIGIBILITY:
Inclusion Criteria:

* All SVR study cohort members will be contacted to assess for vital status. Transplant free survivors will be approached to participate in the in-person assessment.

Exclusion Criteria:

* Patients who have undergone cardiac transplantation or biventricular conversion from all outcomes other than vital status.
* Those with pacemakers will be excluded from the CMR, and patients <130 cm in height will be excluded from the exercise test.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All SVR study cohort members will be contacted to assess for vital status. Transplant free survivors will be approached to participate in the in-person assessment.
Sampling Method: Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2015-06; Primary Completion 2020-10 (Actual); Study Completion 2025-12 (Estimated)

REFERENCES:
- [Derived] Miller TA, Sharma B, Gongwer R, Trachtenberg FL, Newburger JW, Goldberg CS, Gustafson KE, Gaynor JW, Votava-Smith JK, Lambert LM, Sananes R, Kral MC, Tsang R, Heinrich KP, Cnota J, Shah A, Ilardi D; Pediatric Heart Network Investigators. Neurodevelopmental Outcomes in Early Adolescence: The Pediatric Heart Network's Single Ventricle Reconstruction Trial. Circulation. 2025 Oct 28;152(17):1246-1261. doi: 10.1161/CIRCULATIONAHA.125.074523. Epub 2025 Jul 17. PMID 40671650

RESULTS

PARTICIPANT FLOW:
Groups:
- mBTTS: Blalock Taussig Thomas shunt at Norwood
- RVPAS: right-ventricular-to-pulmonary-artery shunt at Norwood
Period: Overall Study
Arm/Group | mBTTS | RVPAS
Started | 109 | 128
Completed | 109 | 128
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | mBTTS | RVPAS | Total
Number analyzed (Participants) | 109 | 128 | 237
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 109 | 128 | 237
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 46 | 93
  Male | 62 | 82 | 144
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 27 | 41
  Not Hispanic or Latino | 95 | 100 | 195
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 95 | 106 | 201
  Non-White | 13 | 21 | 34
  Missing | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: RVEF at 10-12 Years on MRI
Description: RV ejection fraction (RVEF) at 10-12 years, as measured by cardiac magnetic resonance (CMR).
Time Frame: assessed between 10-12 years of age, an average of 53.2 days from consent
Population: participants who underwent cardiac MRI
Measure: Mean (Standard Deviation); unit: percentage of blood pumped
Arm/Group | mBTTS | RVPAS
Number analyzed (Participants) | 75 | 90
percentage of blood pumped | 52 (7.4) | 51 (9.6)

2. Secondary Outcome: Death or Cardiac Transplantation
Description: The incidence of death or cardiac transplantation between those randomized to receive a RVPAS vs. a MBTS at the time of the Norwood operation.
Time Frame: 11 years ± 1 year to 16 years
Reporting Status: Not Posted

3. Secondary Outcome: The Exercise Tolerance Between Those Randomized to a RVPAS vs. a MBTS.
Description: Exercise capacity: Maximal Oxygen Consumption (VO2max), maximal work rate, and anaerobic threshold
Time Frame: 11 years ± 1 year to 16 years
Reporting Status: Not Posted

4. Secondary Outcome: Atrial and Ventricular Arrhythmias
Description: The incidence of arrhythmias between those randomized to a RVPAS vs. a MBTS.
Time Frame: 11 years ± 1 year to 16 years
Reporting Status: Not Posted

5. Secondary Outcome: The Neurodevelopmental Outcomes at 11 Years of Age in Those Randomized to a RVPAS vs. a MBTS
Description: Achievement, as measured by the Wechsler Individual Achievement Tests (WIAT) (Math and Reading); Intelligence, as measured by the Wechsler Intelligence Scale for Children (WISC); Other domains of neurodevelopmental function including assessment of language, executive function, visual spatial skills, motor function, memory, social skills, behavior, health-related quality of life (HRQoL) and adaptive function.
Time Frame: 11 years ± 1 year
Reporting Status: Not Posted

6. Secondary Outcome: Risk Stratification Models
Description: Develop risk stratification models for 1) cardiac outcomes, 2) transplant-free survival, and 3) neurodevelopmental outcomes.
Time Frame: 11 years ± 1 year to 16 years
Reporting Status: Not Posted

7. Secondary Outcome: Biospecimens
Description: Collect specimens from subjects and their parents to further develop the biologic specimen repository.
Time Frame: 11 years ± 1 year to 16 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: through study completion, an average of 5.3 years from consent
Description: through study completion
Arm/Group | mBTTS | RVPAS
All-Cause Mortality (participants affected / at risk) | 3/109 | 3/128
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/128
Other Adverse Events (participants affected / at risk) | 0/109 | 0/128

LIMITATIONS AND CAVEATS:
We cannot exclude enrollment bias or survival bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-28): https://cdn.clinicaltrials.gov/large-docs/31/NCT02455531/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-28): https://cdn.clinicaltrials.gov/large-docs/31/NCT02455531/ICF_001.pdf